CLINICAL TRIAL: NCT00443794
Title: A Randomized Double Blind Controlled Trial of the Efficacy and Safety of POLYCAP (Quintapill)Versus Its Components in Subjects With at Least One Additional Cardiovascular Risk Factor
Brief Title: The Indian POLYCAP Study (TIPS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. John's Research Institute (Other)
Collaborators: Cadila Pharnmaceuticals (Industry); Population Health Research Institute (Other)
Responsible Party: Project Director, The Indian Polycap Study Steering Comittee., Division of Clinical Trials, St. John's Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Rx-Medical-CVS-06-01
Record Dates: First submitted 2007-02-14; First posted 2007-03-06 (Estimated); Last update posted 2010-09-23 (Estimated); Status verified 2010-09

CONDITIONS: Cardiovascular Diseases
Keywords: POLYCAP, Primary Prevention,CVD
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Thiazides; Ramipril; Atenolol; Simvastatin; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- 1, POLYCAP (Experimental): Combination of 3 anti hypertensives, lipid lowering agent and anti platelet agent
  Interventions: Drug: POLYCAP
- 2 B (Active Comparator): Diuretic antihypertensive
  Interventions: Drug: Thiazides
- 3 C (Active Comparator): Thiazide plus Angiotensis converting enzyme inhibitor - combination antihypertensive.
  Interventions: Drug: Ramipril with Thiazide
- 4 D (Active Comparator): Diuretic with Beta blocker combination antihypertensive
  Interventions: Drug: Thiazide plus atenolol
- 5, E (Active Comparator): ACE inhibitor plus Beta blocker combination antihypertensive
  Interventions: Drug: Ramipril plus atenolol
- 6, F (Active Comparator): Combination antihypertensive of ACE inhibitor, diuretic and beta blocker
  Interventions: Drug: Ramipril plus atenolol plus thiazide
- 7,G (Active Comparator): Combination of ACE inhibitor, betablocker, diuretic and Antiplatelet
  Interventions: Drug: Thiazide + Ramipril+Atenolol+Aspirin
- 8,H (Active Comparator): Lipid lowering agent
  Interventions: Drug: Simvastatin
- 9,A (Active Comparator): Antiplatelet
  Interventions: Drug: aspirin

INTERVENTIONS:
Drug: Thiazides — Capsule (blinded) oral administration once daily for 12 weeks
  Arms: 2 B
Drug: Ramipril with Thiazide — Capsule (blinded) oral administration 12 weeks
  Arms: 3 C
Drug: Thiazide plus atenolol — Caspule (blinded) for oral administration once daily for 12 weeks
  Arms: 4 D
Drug: Ramipril plus atenolol — Capsule ( blinded) for oral administration once daily for 12 weeks
  Arms: 5, E
Drug: Ramipril plus atenolol plus thiazide — Capsule (blinded) for oral administration once daily for 12 weeeks
  Arms: 6, F
Drug: POLYCAP — Capsule for Oral Administration once daily for 12 weeks
  Other Names: Quintapill(R)
  Arms: 1, POLYCAP
Drug: Thiazide + Ramipril+Atenolol+Aspirin — Capsule (Blinded) for oral administration once daily for 12 weeks
  Arms: 7,G
Drug: Simvastatin — Capsule (Blinded) for oral administration once daily for 12 weeks
  Arms: 8,H
Drug: aspirin — capsule (Blinded) for oral administration once daily for 12 weeks
  Arms: 9,A

SUMMARY:
STUDY TITLE A randomized double-blind controlled trial of the efficacy and safety of the POLYCAP® versus its components in subjects aged 45 to 80 years of age with at least one additional cardiovascular risk factor.

STUDY OBJECTIVES This study is designed to assess the efficacy and safety of the POLYCAP®, a fixed dose combinationcontaining 5 drugs (an antiplatelet drug; 3 blood pressure lowering agents, a beta blocker, an ACE inhibitor, a diuretic and a statin.

STUDY DESIGN

Randomized controlled double-blind trial of the POLYCAP® versus its components in eight formulations.

STUDY POPULATION Subjects between 45 and 80 years of age, with at least one additional CVD risk factor.

INVESTIGATIONAL PRODUCTS Composition POLYCAP® and its comparators FOLLOW UP The total duration of follow up will be 4 months, from the start of study medication.. Subjects will take study medication for 3 months. There will be a final follow up visit 1 month after stopping the study medication.

There will be five follow up visits, the first 7 - 10 days after starting study medication and thereafter monthly visits for 4 months. Subjects taking any of the study medications prior to enrolment will have one or more additional visits during a defined wash out and before enrolment.

OUTCOME MEASURES Mean difference of change in BP, LDL and urinary thromboxane at the end of the three month period.

STATISTICAL ISSUES Non-inferiority evaluation of the POLYCAP in modifying BP, lipids and platelet activity [as measured by urinary thromboxane] when compared with its different components in eight different formulations.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 80 years
* At least any one of the following CVD risk factors:

  * Stable type 2 diabetes mellitus or
  * Hypertension or
  * Current smoker or
  * A waist to hip ratio > 0.85 for women and >0.9 for men or
  * Elevated lipids.
* Informed consent.

Exclusion Criteria:

* On any of the study medications,
* Uncontrolled blood pressure,
* Symptomatic hypotension,
* Any clear indication or a contraindication to the use of any of the study medications,
* History of coronary/cerebrovascular events,
* Pregnancy or lactating or women of child-bearing potential with inadequate contraception and / or an inability to attend follow up visits.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2050 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Reduction in blood Pressure | 12 weeks
reduction in Heart Rate | 12 weeks
modify lipids | 12 weeks

SECONDARY OUTCOMES:
Platelet aggregation | 12 weks

CONTACTS AND LOCATIONS:
Overall Officials: Prem Pais, MD Medicinie, Study Chair — Dean, Professor of Medicine, St Johns Medical College, Head Division of Clinical Trials St John's Research Institute, Bangalore, India; Denis Xavier, MD Pharmac, Study Director — HOPE Research Scholar, Department of Medicine, PHRI, McMaster University, Hamilton, ON, Canada,; Salim Yusuf, DPhil,FRCPC,FRSC, Study Chair — Director, Population Health Research Institute, Mc Master University, Hamilton, ON, CANADA
Locations (54):
- India (54):
  - Aditya nursing Home, Adoni, Andhra Pradesh
  - Gowri Gopal Nursing Home, Adoni, Andhra Pradesh
  - Apollo Hospital, Hyderabad, Andhra Pradesh
  - Care Hospital, Banjarahills, Hyderabad, Andhra Pradesh
  - Care Hospital, Nampalli, Hyderabad, Andhra Pradesh
  - Durga Bai Deshmuk Hospital, Hyderabad, Andhra Pradesh
  - Global hospital, Hyderabad, Andhra Pradesh
  - Mahavir Hospital, Hyderabad, Andhra Pradesh
  - Vijaya Durga Cardiac Centre, Kurnool, Andhra Pradesh
  - Vijaya Hospital, Kurnool, Andhra Pradesh
  - Care Hospital, Secunderabad, Andhra Pradesh
  - Krishna Institute of Medical Sciences, Secunderabad, Andhra Pradesh
  - Care Hospital, Visakhapatnam, Andhra Pradesh
  - Care Cardiovascular Consultant, Ahmedabad, Gujarat
  - V S hospital, Ahmedabad, Gujarat
  - Dev Hospital and ICU, Vadodara, Gujarat
  - ST JOHN'S MEDICAL COLLEGE HOSPITAL, Dept of Cardiology, Bangalore, Karnataka
  - St John'S Medical College Hospital, Department of Medicine, Bangalore, Karnataka
  - Mahaveer Jain Hospital, Bangalore, Karnataka
  - Workhardt Hospital, Bangalore, Karnataka
  - Belgaum Diabetes, Belagavi, Karnataka
  - Vikaram Hospital and Health Care, Mysore, Karnataka
  - Nanjappa Hospital, Shimoga, Karnataka
  - Baby Memorial Hospital, Calicut, Kerala
  - Amrita Institute of medical Science, Kochi, Kerala
  - West Fort Hospital, Thrissur, Kerala
  - Kerala Institute of Medical sciences, Trivandrum, Kerala
  - Apex Research Center and Hospital, Bhopal, Madhya Pradesh
  - MGM, Indore, Madhya Pradesh
  - Bhatia Hospital, Mumbai, Maharashtra
  - C H L Apollo Hospital, Mumbai, Maharashtra
  - Health Harmony Hospital, Mumbai, Maharashtra
  - Avanti Institute of Cardiology, Nagpur, Maharashtra
  - Cresent Hospital and Research center, Nagpur, Maharashtra
  - Poona Hospital, Pune, Maharashtra
  - Mahatma Gandhi Institute of Medical Sciences, Wardha, Maharashtra
  - Sri Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Fortis Hospital, Noida, National Capital Territory of Delhi
  - Sidhu Hospital, Ludhiana, Punjab
  - Sadbhavana Heart Institute, Patiāla, Punjab
  - S P Medical College, Bikaner, Rajasthan
  - Monilek Hospital, Jaipur, Rajasthan
  - Tongia Heart Hospital, Jaipur, Rajasthan
  - Bethesda Hospital, Ambur, Tamil Nadu
  - Frontier Lifeline, Chennai, Tamil Nadu
  - Madras Diabetic Research Foundation, Chennai, Tamil Nadu
  - Rajamuthaiah Hospital, Annamalianagar, Chennai, Tamil Nadu
  - Sri Ramachandra Hospital, Chennai, Tamil Nadu
  - PSG Hospital, Coimbatore, Tamil Nadu
  - Ramakrishna Nursing Home, Trichy, Tamil Nadu
  - Christian Medical College Hospital, Vellore, Tamil Nadu
  - King George Hospital, Lucknow, Uttar Pradesh
  - Sanjay Gandhi PGMI, Lucknow, Uttar Pradesh
  - Peerless Hospital and BK Roy esearch Center, Kolkata, West Bengal

REFERENCES:
- [Background] Indian Polycap Study (TIPS); Yusuf S, Pais P, Afzal R, Xavier D, Teo K, Eikelboom J, Sigamani A, Mohan V, Gupta R, Thomas N. Effects of a polypill (Polycap) on risk factors in middle-aged individuals without cardiovascular disease (TIPS): a phase II, double-blind, randomised trial. Lancet. 2009 Apr 18;373(9672):1341-51. doi: 10.1016/S0140-6736(09)60611-5. Epub 2009 Mar 30. PMID 19339045
- [Derived] Xavier D, Pais P, Sigamani A, Pogue J, Afzal R, Yusuf S; Indian Polycap Study (TIPS) Investigators. The need to test the theories behind the Polypill: rationale behind the Indian Polycap Study. Nat Clin Pract Cardiovasc Med. 2009 Feb;6(2):96-7. doi: 10.1038/ncpcardio1438. Epub 2008 Dec 23. No abstract available. PMID 19104516
- See also: Division of Clinical Trials , St John's Research Institute, Website — http://www.sjri.res.in
- See also: Cadila Pharmaceuticals — http://www.cadilapharma.com